CLINICAL TRIAL: NCT03013244
Title: A Randomized Controlled Trial of The Body Project: More Than Muscles for Males With Body Dissatisfaction
Brief Title: Reducing Eating Disorder Risk Factors Among College-Aged Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015.17069
Record Dates: First submitted 2016-12-20; First posted 2017-01-06 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-12

CONDITIONS: Eating Disorder
Keywords: prevention; eating disorder; men; intervention; muscle dysmorphia; peer-led
MeSH Terms: conditions — Feeding and Eating Disorders; Multiple Endocrine Neoplasia Type 1

ARMS (2):
- Waitlist Control (No Intervention): Participants in this condition completed assessments at baseline, 1 week, and 5 weeks.
- The Body Project: More Than Muscles (Experimental): Participants in this condition competed the 2-session dissonance-based eating disorder prevention protocol (2 hours per session).
  Interventions: Behavioral: The Body Project: More Than Muscles

INTERVENTIONS:
Behavioral: The Body Project: More Than Muscles — Participants complete a variety of activities designed to counter internalization of the lean, muscular body ideal for men.
  Arms: The Body Project: More Than Muscles

SUMMARY:
The purpose of the present study was to investigate the acceptability and efficacy of a cognitive dissonance-based (DB) intervention in reducing eating disorder and muscle dysmorphia risk factors in men with body dissatisfaction. The investigators hypothesized that the program would reduce eating disorder risk factors to a greater degree compared to wait list control and that these effects would be maintained at 1 month follow-up.

DETAILED DESCRIPTION:
BACKGROUND & PURPOSE The current project sought to examine the acceptability and efficacy of a cognitive dissonance-based (DB) eating disorder prevention program for college-aged men with body image concerns. Eating disorders represent a public health problem for which efficacious, disseminable treatments largely remain unknown, particularly for males. Epidemiological data support the increasing prevalence of eating disorders and body image concerns among men; however, few programs have been developed to address concerns relevant to men, and many men feel uncomfortable in programs that identify eating disorders as a "female" problem. Given that eating disorders are particularly difficult to treat, disseminable interventions that can target high-risk groups prior to eating disorder onset may be the best way to reduce the public health burden associated with eating disorders. As body image concerns represent the most potent and consistent risk factor for developing eating disorders in males and females, men with body image concerns represent one such high-risk, but underserved, group.

Recent prevention research has used DB principles to challenge thin-ideal internalization to decrease the likelihood of developing an eating disorder in female youth. Additionally, the investigators recently adapted and evaluated a DB program for gay males (The PRIDE Body Project), who represent another high-risk group among men. Dissonance theory states that when individuals engage in counter-attitudinal behavior they experience psychological discomfort, leading them to alter their attitudes to be congruent with their behavior. Several studies have supported the efficacy of DB programs in reducing eating disorder risk among females and results from The PRIDE Body Project extends the efficacy of these programs to gay males. These DB interventions have utilized peer co-leaders, capitalizing on the importance of peer influences on eating behaviors among college-aged females and males.

To date, other than The PRIDE Body Project, no studies have examined eating disorder prevention interventions for high-risk groups of males. Notably, the success of The PRIDE Body Project and several lines of research support that adapting a DB program may also be helpful in reducing eating disorder risk among young men with body image concerns. First, internalization of the mesomorphic ideal plays a central role in risk for developing eating pathology in males. Thus, an intervention targeting internalization of this body ideal may be particularly helpful for males. Second, studies support that peers influence body dissatisfaction and disordered eating in males concurrently and prospectively through socialization. This suggests that men, regardless of sexual orientation, may benefit from a peer-led DB program to address body image concerns. This work could fill a critical gap in the care provided to a growing demographic among those who suffer from eating disorders.

Thus, the aim of the present study was to determine the acceptability and efficacy of adapting a cognitive DB intervention for use in college-aged men with body image concerns. 112 men with body image concerns were recruited to participate in a randomized controlled trial (RCT), in which they were randomized into either a DB intervention (n=52) or wait list control (WL) condition (n=60).

The investigators hypothesized that: (1) The men in the DB group would show significantly greater reductions on all measures compared to men in the WL group; and (2) Differences between groups would be maintained at 4-week follow-up.

DESIGN Participants Participants (n=112) were recruited through introductory and upper division psychology classes at Florida State University (FSU), through the psychology research participant pool, and advertisements around the campus and local community. Based on retention rates in The PRIDE Body Project, the investigators estimated a 75% retention rate. Analyses support that the expected sample size should provide sufficient power to detect group differences, based on effect sizes from previous DB studies.

Procedure All participants first completed an eligibility phone screen to determine whether they met study eligibility criteria. Participants who qualified for and were interested in participating in the study were directed to complete the online consent form.

This intervention was adapted from a two-session DB intervention that the investigators developed for gay men, which was originally adapted for women to address risk factors specific to males with body image concerns, regardless of sexual orientation. Participants completed baseline measures assessing eating disorder and muscle dysmorphia risk factors, which were selected based on demonstrated reliability and validity in previous studies, particularly for use in men.

The two, 2-hour intervention sessions were spaced one week apart. Intervention groups included 4-10 members each and took place at the FSU psychology building. The investigator and an undergraduate peer co-leader facilitated all intervention groups. During Session 1, participants: (a) defined the male "body-ideal", (b) discussed the origin/perpetuation of the "body-ideal", (c) brainstormed costs of pursuing the "ideal", (d) participated in verbal challenges countering the "body-ideal" message, and (e) were assigned homework assignments. In Session 2 participants: (a) reviewed homework, (b) engaged in role plays to counter pursuit of the "body-ideal" (c) discussed ways to challenge and avoid negative "body talk" (d) listed ways to resist pressures to pursue this ideal both individually and at the university level (termed "body activism") and (e) selected an exit exercise to practice positive body talk. All intervention sessions were audiotaped to ensure facilitator adherence to the protocol.

Baseline measures were repeated for both conditions immediately post-intervention/after a one-week interval and 4-weeks post-intervention/after a five-week interval, to assess immediate and longer-term effects.

Data Analytic Plan The data analytic approach utilized hierarchical linear modeling (HLM), to control for repeated assessments of participants nested within groups.

ELIGIBILITY:
Inclusion Criteria:

* male
* do not meet criteria for an eating disorder (based on phone screen interview)
* endorse body image concerns
* 18 years -30 years
* agree to participate in a positive body image program.

Exclusion Criteria:

* Individuals under 18 years of age
* Individuals who do not meet criterion a, b, c, or d (as outlined in the inclusion criteria)
* Individuals who meet full criteria for an eating disorder based on responses on the phone screen

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2014-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Eating Disorder Examination Questionnaire - Bulimic Symptoms Composite | change from baseline to post-intervention (1 week)
Sociocultural Attitudes Towards Appearance Questionnaire-3 - Internalization General subscale | change from baseline to post-intervention (1 week)
Eating Disorder Examination-Questionnaire Restraint Subscale | change from baseline to post-intervention (1 week)
Male Body Attitudes Scale | change from baseline to post-intervention (1 week)
  The investigators examined the Muscularity and Body Fat subscales for this study
Drive for Muscularity Scale | change from baseline to post-intervention (1 week)
Muscle Dysmorphia Disorder Inventory | change from baseline to post-intervention (1 week)

SECONDARY OUTCOMES:
Eating Disorder Examination Questionnaire - Bulimic Symptoms Composite | change from baseline to follow-up (5 weeks)
Sociocultural Attitudes Towards Appearance Questionnaire-3 - Internalization General subscale | change from baseline to follow-up (5 weeks)
Eating Disorder Examination-Questionnaire Restraint Subscale | change from baseline to follow-up (5 weeks)
Male Body Attitudes Scale | change from baseline to follow-up (5 weeks)
  The investigators examined the Muscularity and Body Fat subscales for this study
Drive for Muscularity Scale | change from baseline to follow-up (5 weeks)
Muscle Dysmorphia Disorder Inventory | change from baseline to follow-up (5 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela K Keel, PhD, Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No